CLINICAL TRIAL: NCT06874985
Title: Effectiveness and Impact of the Lived Experience Cancer Awareness Campaign on Participation in the Existing Cancer Screening Programs [Oral, Breast and Cervical] Among the Rural Population in Villupuram District, Tamil Nadu
Brief Title: Effectiveness and Impact of the Lived Experience Cancer Awareness Campaign on Screening Participation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: International Agency for Research on Cancer (Other)
Collaborators: Adyar Cancer Institute, WIA, Chenni, India (Unknown); Department of Public Health and Preventive Medicine (DPH & PM), Chennai, India (Unknown)
Responsible Party: Principal Investigator, Partha Basu, Dr, International Agency for Research on Cancer
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IEC 22-05; MR/W023903/1 (Other Grant/Funding Number: Medical Research Council (MRC))
Record Dates: First submitted 2025-02-28; First posted 2025-03-13 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Cervical Cancers; Breast Cancer; Oral Cancer
Keywords: Lived Experience Communication Campaign; Randomised control trial; Cancer screening; Public Health intervention; Access Cancer Care India
MeSH Terms: conditions — Uterine Cervical Neoplasms; Breast Neoplasms; Mouth Neoplasms

STUDY DESIGN:
Intervention Model Description: Since cluster or individual randomization was not feasible due to the risk of contamination, a simple randomization strategy was employed at the block-level. A coin flip [doe by the investigator team at IARC] identified which block would receive the intervention (Mailam) and which would serve as the control (Vanur). However, all the baseline characteristics and demographics will be collected from both the participants in both villages and would be compared to ensure
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Participants in the selected villages will be shown a two-minute video developed specifically for the Lived Experience Communication Campaign in addition to usual awareness they receive for cancer screening mobilisation. The video will feature personal narratives from cancer survivors and local leaders emphasizing the importance of early detection and screening.
  Interventions: Behavioral: Lived experience video campaign
- Control arm (No Intervention): Participants will receive standard cancer awareness campaigns conducted by community health workers as per existing healthcare practices. No additional materials or interventions will be provided beyond routine awareness programs.

INTERVENTIONS:
Behavioral: Lived experience video campaign — Participants in the selected villages will be shown a two-minute video developed specifically for the Lived Experience Communication Campaign in addition to usual awareness they receive for cancer screening mobilisation. The video will feature personal narratives from cancer survivors and local leaders emphasizing the importance of early detection and screening.
  Arms: Intervention arm

SUMMARY:
This study will be conducted as a parallel-arm, open-label, randomized controlled trial (RCT) to evaluate the effectiveness and impact of the Lived Experience Communication Campaign (LECC) on cancer screening participation rates [oral, breast and cervical cancer] compared to the usual standard awareness campaign across selected rural population in Villupuram district, Tamil Nadu.

DETAILED DESCRIPTION:
The Access Cancer Care India (ACCI) project is aimed at designing and evaluating an evidence-based multi-level strategy tailored to the local health system to enhance access to early detection and care continuum for oral, breast, and cervical cancers among rural populations in India, who are socioeconomically disadvantaged and vulnerable to huge inequity in cancer care.

Pre-intervention phase:

The pre-intervention assessment was conducted in four blocks (Vanur, Mailam, Vikravandi, Kanai) in Viluppuram District, Tamil Nadu, between August 2023 and July 2024 to understand the barriers and challenges rural men and women face in accessing cancer early detection care continuum using various methods.

1. Questionnaire survey of breast, cervical, and oral cancer patients and the general population
2. Focus group discussions with the general population and community health workers
3. In-depth interviews with key informants
4. Capacity assessment The results of the preintervention highlighted that fear, stigma, limited accessibility to screening, miscommunication and lack of family support were vital barriers that influenced cancer care access in Tamil Nadu. Thus, we decided to design and implement evidence based cultural relevant intervention, pilot test and evaluate them. In order to target the component of fear, stigma and accessibility issues, we decided to design and implement a Lived life communication campaign and test it as an RCT across selected blocks of Tamil Nadu. The rationale for proposing a parallel-arm RCT for this intervention is to assess its effectiveness specifically within the Indian context. While the "lived experience" campaign has been successfully implemented in other Asian populations, its impact in India remains untested. A parallel-arm RCT design enables comparison across the intervention and control arm on specific screening program outcomes. This approach ensures a comprehensive assessment of the intervention's effectiveness in improving screening uptake among the target population. The findings will provide robust evidence to either validate or improve the intervention, tailoring it to the unique needs of the Indian setting. This study evaluates the effectiveness of the Lived Experience Communication Campaign (LECC) in increasing participation in cancer screening programs for oral, breast, and cervical cancer among rural populations in Villupuram district, Tamil Nadu. Conducted as a parallel-arm, open-label, randomized controlled trial (RCT), the study compares LECC to standard awareness campaigns. Randomisation was at the level of the block using cointoss, where Mailam block serves as the intervention site, while Vanur block serves as the control. Eligible participants (men and women aged 30-59 years without prior cancer diagnoses or recent screenings) will be randomly selected using systematic sampling. The intervention comprises a culturally relevant two-minute awareness video featuring personal survivor narratives, delivered door-to-door by community health workers. Standard awareness campaigns are conducted in the control arm. Baseline data on cancer screening participation is collected from healthcare records. Follow-up assessments are conducted monthly for six months, measuring screening participation rates and other program indicators. Evaluation follows the RE-AIM framework, examining effectiveness, feasibility, and acceptability. Results will inform future policy decisions on implementing lived experience campaigns to enhance cancer screening uptake in India.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 30-59 years
* No prior diagnosis of cervical, breast, or oral cancer.
* Have not undergone screening for the above cancers in the last 1 year
* Provide informed consent to participate

Exclusion Criteria:

* Individuals with a previous history of any cancer
* Individuals with severe cognitive impairments that prevent comprehension of study materials
* Participants unwilling to provide informed consent

Ages: 30 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1120 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Screening Participation Rate | 1 month after the participation
  The proportion of eligible participants who visited a healthcare center for cervical, breast, or oral cancer screening within one month of the intervention (or usual care in the control group).
Invitation coverage in both arms | 6 months
  The proportion of eligible individuals living in the intervention and control villages covered through invitations for cancer screening.
Examination coverage in both arms | 6 months
  The proportion of individuals eligible for screening who participated in the screening program.
Further assessment coverage in both arm | 6 months
  The proportion of individuals who participated in the cancer screening program requiring further assessment.
Detection of cancers in both arms | 6 months
  The proportion of individuals eligible for screening who are diagnosed with cancers.
Treatment referral in both arms | 6 months
  The proportion of individuals eligible for screening who are referred for treatment to higher centres.

SECONDARY OUTCOMES:
Implementation research outcomes - Reach | 6 months
  Proportion of eligible men and women who received the intervention.
Implementation research outcomes - Effectiveness | 6 months
  Proportion of eligible men and women who agreed to participate in the existing cancer screening program.
Implementation research outcomes - Acceptability | 6 months
  Proportion of eligible men and women who find the intervention (Lived experience campaign video) to be acceptable.

CONTACTS AND LOCATIONS:
Overall Officials: T.S. Selvavinayagam, MD, Principal Investigator — Department of Public Health and Preventive Medicine; Jerard Maria Selvam, Principal Investigator — National Health Mission-Tamil Nadu; K. Krishnaraj, Principal Investigator — Department of Public Health and Preventive Medicine; Vidhya Viswanathan, Principal Investigator — Department of Public Health and Preventive Medicine; N.V. Vani, PhD, Principal Investigator — Cancer Institute (WIA), Chennai; R. Swaminathan, PhD, Principal Investigator — Cancer Institute (WIA), Chennai, India
Locations (1):
- Adyar cancer institute, Chennai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: Undecided